CLINICAL TRIAL: NCT05789654
Title: Accuracy of PADUA PREDICTION SCORE in Thromboembolic Risk Stratification of Cirrhotic Patients Hospitalized in a Non-surgical Environment
Brief Title: PADUA PREDICTION SCORE in Cirrhotic Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Zocco Maria Assunta, Prof, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 3394
Record Dates: First submitted 2023-03-16; First posted 2023-03-29 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-08

CONDITIONS: Portal Thrombosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Primary objective: to evaluate the predictive role of Prediction Score on the risk of developing venous thromboembolism in patients with liver cirrhosis admitted to non-surgical wards.

Secondary objectives:

* To estimate the prevalence and incidence of venous thromboembolism in patients with liver cirrhosis admitted to non-surgical wards
* To calculate the prevalence in the same subset of patients of major bleeding (defined as bleeding resulting in the patient's death, a drop in hemoglobin > 2g/L, the need to transfuse > 2 units of packed red blood cells or bleeding into a critical organ/space including the intracranial, retroperitoneal, intraocular, adrenal, spinal, pericardial districts) related to the application or not of thromboprophylaxis measures (pharmacological and mechanical) Study design: The study is single center and it will be divided into two parts, a first retrospective part and a second prospective case control study.

Methods: adult patients with liver cirrhosis admitted in Internal Medicine and Gastroenterology Unit of Policlinico Agostino Gemelli will be enrolled in the prospective study. For the retrospective part of the study, data about cirrhotic patients hospitalized in non-surgical departments of Policlinico Agostino Gemelli will be collected. Exclusion criteria will be hospitalization in surgical wards or intensive care units, patients with active bleeding at the time of admission, patients hospitalized for liver transplantation, anticoagulant therapy at therapeutic dosage at the time of admission for indications other than liver cirrhosis (e.g. personal history of thromboembolic events, atrial fibrillation/flutter or mechanical heart valves), contraindications to anticoagulant prophylaxis (recent or ongoing bleeding, creatinine clearance assessed by EPI-CKD method < 15 ml/min, platelet count < 50 x 10^9/L), patients hospitalized as elective regimen to perform invasive procedures that contraindicate anticoagulant prophylaxis (e.g. liver biopsy, local treatment of liver neoplasms, ligation of oesophageal varices), double antiplatelet therapy, pregnancy

ELIGIBILITY:
Inclusion Criteria:

* written informed consent
* age more than 18 years old
* diagnosis of liver cirrhosis
* hospitalization in a medical department

Exclusion Criteria:

* pregnancy
* ongoing double anticoagulation or double antiplatelet therapy at the moment of hospitalization
* controindications to anticoagulation therapy
* hospitalization in surgical environnment

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: adult cirrothic patients hospitalized in non surgical environnment
Sampling Method: Non-Probability Sample
Enrollment: 132 (Estimated)
Dates: Start 2020-09-10 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
predicting venous thromboembolic risk in liver cirrhosis | 12 months
  evaluating Padua Prediction Score role in predicting venous thromboembolic risk in liver cirrhosis

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Gemelli IRCCS, Roma, Italy